CLINICAL TRIAL: NCT07382141
Title: Early Identification of Cardivascular Damage Induced by Chemotherapy and Antineoplastic Treatments in Pediatric Age
Acronym: PREDICT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRE.D.I.C.T.
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiotoxicity
Keywords: cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Parameters of vascular stiffness — VICORDER© is a noninvasive, quick and painless technique to be able to assess vascular elasticity and consists of placing a few sphygmomanometers (the same ones used to measure blood pressure) for a few minutes

SUMMARY:
To test whether the implementation of new diagnostic techniques (ultrasonography, speckle tracking, vascular stiffness study, cardiac MRI, and histologic studies) allows in CAYA (Childern, Adolescents, and Young Adults) cancer survivors a more sensitive and earlier identification of cardiovascular damage resulting from antineoplastic therapy that develops either acutely or remotely after completion of antineoplastic therapy.

DETAILED DESCRIPTION:
Cardiovascular system is among the main target organs of toxicity of some antineoplastic treatments. Pretreatment cardiotoxicity risk stratification and timing tailored to patient needs are strategies recognized in cardiology but not yet well validated in the pediatric population. Currently, follow-up of the pediatric patient diagnosed with oncologic disease involves serious cardiologic evaluation, independent of cardiovascular risk factors and focused on recognition of left ventricular systolic dysfunction. The use of new diagnostic methods to study the pediatric patient exposed to antineoplastic therapy and the personalization of follow-up on the basis of pretreatment cardiovascular risk could allow early identification of cardiotoxic damage and thus prevent its progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of oncological pathology and need for antineoplastic treatment

Exclusion Criteria:

* None

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular events in CAYA cancer survivors during treatment and follow-up | From initiation of antineoplastic therapy up to 12 months post-therapy
  Number of cardiovascular events, defined according to ESC 2022 guidelines (Eur Heart J. 2022;43:4229-4361), detected during treatment and follow-up. Time to occurrence of events will be measured relative to pre-treatment evaluation.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - IRCCS - AOU di Bologna -Policlinico di Sant'Orsola UOC Pediatria, Bologna, Bologna
  - IRCCS AOU di Bologna -Policlinico di Sant'Orsola UO Cardiochirurgia pediatrica e dell'età evolutiva, Bologna, Bologna
  - IRCCS AOU di Bologna -Policlinico di Sant'Orsola UO Oncoematologia Pediatrica, Bologna, Bologna
  - IRCCS AOU di Bologna Policlinico di Sant'Orsola UO Cardiologia Pediatria e dell'età evolutiva, Bologna, Bologna
  - IRCCS AOU di Bologna Policlinico di Sant'Orsola UO Radiologia, sezione Cardio-Toraco-Vascolare, Bologna, Bologna